CLINICAL TRIAL: NCT07031557
Title: Osteoporosis Project in Pregnancy and Lactation (POI)
Brief Title: Pregnancy and Lactation- Associated Osteoporosis
Acronym: POI
Status: Active, not recruiting | Type: Observational
Sponsor: Parma University Hospital (Other)
Responsible Party: Principal Investigator, Tullio Ghi, Principal Investigator, Medical Doctor, Professor of Obstetrics and Gynecology, Parma University Hospital
Other Study IDs: POI
Record Dates: First submitted 2025-03-03; First posted 2025-06-22 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-06

CONDITIONS: Osteoporosis and Fracture Risk in Pregnant Women
Keywords: Pregnancy-Associated Osteoporosis; REMS
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pregnant and Breastfeeding Women: Participants in this cohort are pregnant women enrolled during their first trimester and followed up through the third trimester and the breastfeeding period. They will undergo a structured assessment of bone health, including completion of
  * two standardized questionnaires, Calcium Intake and Dietary Habits Questionnaire, based on the PREDIMED score to assess adherence to the Mediterranean diet;
  * AFEF Questionnaire (Algorithm for Fracture Risk in Women of Fertile Age), to evaluate clinical, anthropometric, pharmacological and lifestyle risk factors for fragility fractures.
  Additionally, they will use REMS technology to monitor bone health, with periodic evaluations (first trimester, third trimester, and six months postpartum) for bone mineral density (BMD, g/cm²) and Fragility Score (0-100 scale) measurements.
  Interventions: Device: EchoStation Implementing REMS Technology; Other: Nutritional and Fracture Risk Assessment Questionnaires

INTERVENTIONS:
Device: EchoStation Implementing REMS Technology — Ultrasound-based densitometry used for the prevention, diagnosis, and monitoring of bone health status and fracture risk at reference anatomical sites (femur and spine), including all patient categories.
  Other Names: EchoStation (Echolight S.p.A.)
Other: Nutritional and Fracture Risk Assessment Questionnaires — Questionnaires regarding Calcium Intake, dietary habits assessment (Predimed), and Algorithm for Fracture Risk in Women of Childbearing Age (AFEF) developed by the Fragility Fracture Observatory (OFF)

SUMMARY:
Pregnancy-Associated Osteoporosis is a condition characterized by loss of bone mass and fragility fractures during pregnancy or breastfeeding, often due to the increased calcium request from fetus. It typically manifests from the third trimester of pregnancy or in the early months of breastfeeding. Therefore, early diagnosis is crucial to prevent fractures and vertebral collapses.

The study aims to monitor bone mineral density (BMD) and fracture risk in pregnant and breastfeeding women using:

1. Questionnaires on calcium intake, dietary habits (Predimed), and fracture risk (AFEF);
2. Ultrasound densitometry (REMS) in the first and third trimester of pregnancy and during breastfeeding.

ELIGIBILITY:
Inclusion Criteria:

* Signature informed consent
* Willingness to participate in the study and ability to complete the study-related questionnaires
* Women in the first trimester of pregnancy at the time of inclusion in the study
* Age between 18 and 45 years at the time of recruitment in the study
* Absence of secondary osteoporosis (induced by diseases or medication use)
* Absence of current or past conditions that could potentially interfere with bone metabolism (e.g., thyroid, kidney, or liver diseases)
* Women of normal weight or with class I obesity (BMI between 18,5 and 34)

Exclusion Criteria:

* Absence of informed consent
* Low compliance and/or inability to complete the study-related questionnaires
* Women not beyond the first trimester of pregnancy and pregnancy-related or pre-existing comorbidities
* Age under 18 or over 45 years
* BMI less than 18.5 or greater than 34

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A cohort of 1230 pregnant women aged 18-45 years and BMI between 18.5 and 34 without secondary osteoporosis and potential pathological conditions that may affect bone health.
Sampling Method: Probability Sample
Enrollment: 1230 (Actual)
Dates: Start 2024-09-09 (Actual); Primary Completion 2025-09-08 (Estimated); Study Completion 2026-09-08 (Estimated)

PRIMARY OUTCOMES:
Calcium- intake Questionnaire | Baseline (First Trimester, ≤12 weeks), Third Trimester (Weeks 28-40), and 6 Months Postpartum
  Daily calcium intake will be estimated using a semi-quantitative dietary questionnaire developed by the Fragility Fracture Observatory (OFF). The questionnaire collects data on the consumption frequency and portion size of calcium-rich foods. Results will be analyzed to determine whether calcium intake meets the physiological needs during pregnancy and breastfeeding.
  There is no predefined score; intake will be expressed in estimated milligrams (mg) of calcium per day based on food composition and reported consumption patterns.
AFEF Questionnaire | Baseline (First Trimester, ≤12 weeks), Third Trimester (Weeks 28-40), and 6 Months Postpartum
  Fracture risk will be assessed through the AFEF (Algorithm for Fracture Risk in Women of Fertile Age) questionnaire developed by the Fragility Fracture Observatory (OFF). The questionnaire is a non-scoring, structured tool collecting detailed information on anthropometrics (e.g., weight and height), personal and family medical history, lifestyle factors (e.g., smoking), and pharmacological treatments before and during pregnancy.
  No numerical score is generated. Risk profiles will be evaluated qualitatively based on the presence or absence of recognized clinical risk factors for fragility fractures.
PREDIMED Score for Mediterranean Diet Adherence | Baseline (First Trimester, ≤12 weeks), Third Trimester (Weeks 28-40), and 6 Months Postpartum
  Adherence to the Mediterranean diet will be assessed using the validated PREDIMED questionnaire, which includes 14 items evaluating dietary habits. Each item is scored as 1 (adherent) or 0 (non-adherent), for a total score ranging from 0 to 14.
  Scores are interpreted as follows: ≤5 = Low adherence, 6-9 = Moderate adherence, ≥10 = High adherence.
  Higher scores indicate better adherence to the Mediterranean diet.

SECONDARY OUTCOMES:
Change in Bone Mineral Density (BMD) at the Proximal Femur Assessed by REMS During Pregnancy and Breastfeeding | Baseline (First Trimester, ≤12 weeks), Third Trimester (Weeks 28-40), and 6 Months Postpartum
  To monitor longitudinal changes in bone structure by measuring Bone Mineral Density (BMD unit g/cm²) using Radiofrequency Echographic Multi Spectrometry (REMS) at the proximal femur. Assessments will occur during the first trimester, third trimester of pregnancy and during breastfeeding. Results will be reported separately for participants stratified into two baseline BMD groups (normal vs. reduced).
Fragility Score (FS) Measured by REMS at the Proximal Femur During Pregnancy and Breastfeeding | Baseline (First Trimester, ≤12 weeks), Third Trimester (Weeks 28-40), and 6 Months Postpartum
  To evaluate the risk factors that lead to variations in bone fragility, through the use of the REMS-based Fragility Score (FS) parameter, identifying the cut-off value for femoral FS specific to pregnant women.
  Unit of Measure of Fragility Score (FS), scale 0-100, where higher FS values represent increased fragility.

CONTACTS AND LOCATIONS:
Locations (1):
- Tullio Ghi, Parma, Italy/Parma, Italy

IPD SHARING:
Plan to Share IPD: No